CLINICAL TRIAL: NCT05033314
Title: THromboprophylaxis In Sickle Cell Disease With Central Venous Catheters (THIS): A Pilot Study
Brief Title: THromboprophylaxis In Sickle Cell Disease With Central Venous Catheters (THIS)
Acronym: THIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to slow recruitment.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-5846.0
Record Dates: First submitted 2021-08-05; First posted 2021-09-02 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease; Central Venous Catheter Thrombosis; Venous Thromboembolism
MeSH Terms: conditions — Anemia, Sickle Cell; Upper Extremity Deep Vein Thrombosis; Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban thromboprophylaxis (Experimental)
  Interventions: Drug: Rivaroxaban 10 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Rivaroxaban 10mg PO daily as thromboprophylaxis
  Other Names: Xarelto 10mg
  Arms: Rivaroxaban thromboprophylaxis
Drug: Placebo — matching placebo daily
  Arms: Placebo

SUMMARY:
Research Question:

In adult SCD patients with CVC, is it feasible and safe to conduct an adequately powered RCT to evaluate the use of rivaroxaban as thromboprophylaxis in this population?

Study Design:

The study is a vanguard pilot double blind multi-centre randomized controlled trial. Participants with SCD and CVC will be randomized to either rivaroxaban 10mg PO daily or placebo for the duration of CVC in situ or for up to one year, whichever is less. After screening (day -7 to day -1), patients will be followed at day 1, months 3 (+/- 15 days), 6 (+/- 15 days), 9 (+/- 15 days), and 12 (+/- 15 days).

Study Objectives:

The primary objective is to estimate the proportion of eligible patients who will enroll into a trial of thromboprophylaxis.

Secondary objectives include (a) document indications for central venous catheter (CVC), (b) summarize duration of CVC insertion prior to enrollment, (c) estimate adherence to the study drug, (d) estimate proportions of participants being compliant with study procedures, and lost to follow up.

Exploratory objectives will assess thrombotic, bleeding, and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age 18 or older)
2. Documented SCD
3. New or pre-existing CVC planned for long term use (at least 6 months)
4. Able to provide written consent

Exclusion Criteria:

1. Contra-indication to prophylactic dose anticoagulation or active bleeding at discretion of treating physician
2. Already on anticoagulation (prophylactic or therapeutic dose) for an indication other than CVC thromboprophylaxis
3. Previous VTE within the past 3 months
4. Pregnant, within 6 weeks post-partum, or active breast feeding
5. Creatinine clearance <30mL/min (as calculated by Cockcroft-Gault equation[67])
6. Acute hepatitis or chronic active hepatitis
7. Cirrhosis with Child-Pugh score B or C
8. Platelet count < 50 x109/L
9. Weight <40kg
10. Uncontrolled HTN (systolic blood pressure > 170mmhg, or diastolic blood pressure> 100mmhg) despite antihypertensive treatment
11. On palliative care
12. On dual antiplatelet therapy, or high dose single agent aspirin > 325mg/day
13. On combined P-glycoprotein and strong cytochrome P450 3A4 inhibitors (including but not limited to ketoconazole and protease inhibitors)
14. On combined P-glycoprotein and strong cytochrome P450 3A4 inducers (including but not limited to rifampin, phenytoin, phenobarbital, carbamazepine, and st. john's wort)
15. Active cancer or treatment for cancer excluding basal cell carcinoma
16. Known allergy to study drug
17. Strong indication for thromboprophylaxis at discretion of treating physician
18. Significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible patients who will enroll into a trial of thromboprophylaxis | 1 year

SECONDARY OUTCOMES:
Document indications for central venous catheter (CVC) | 1 year
Summarize duration of CVC insertion prior to enrollment | 1 year
Estimate adherence to the study drug | 1 year
  1. Adherence: percentage of administered drugs not returned (by pill counting);
  2. Compliance: defined as percentage adherence >80%.
Estimate participants compliance with study procedures, and lost to follow up | 1 year
  Defined as proportion of participant lost to follow up or withdrawn from the study prior to completion of 6 months of treatment

OTHER OUTCOMES:
Venous thromboembolism (VTE) | 1 year
  Proportion of participants with VTE (including CRT, right atrial or ventricular thrombus, proximal DVT, segmental PE, unusual site VTE), and unexplained death in which PE could not be ruled out. CRT is defined to include a proximal vein and must be the same limb as the CVC. Proximal veins include both lower and upper limb, and must include the popliteal or more proximal vein if lower limb, or axillary or more proximal. Unusual site VTE is defined to include cerebral vein thrombosis or splanchnic vein thrombosis. VTE must be objectively confirmed with appropriate imaging modalities.
Major bleeding or clinically relevant non-major bleeding | 1 year
  Defined as per International Society on Thrombosis and Haemostasis (ISTH) criteria
Major bleeding | 1 year
  Defined as per International Society on Thrombosis and Haemostasis (ISTH) criteria
Clinically relevant non-major bleeding | 1 year
  Defined as per International Society on Thrombosis and Haemostasis (ISTH) criteria
Event-free survival | 1 year
  Defined as free from VTE or major bleeding events
Arterial thrombotic events | 1 year
  Including myocardial infarction, ischemic stroke, and systemic embolism
CVC change due to thrombosis or catheter occlusion not amenable to infusion of thrombolytics between study arms | 1 year
  Proportion of participants requiring CVC change due to thrombosis or catheter occlusion not amenable to infusion of thrombolytics
Quality of life using the modified Duke Anticoagulation Satisfaction Scale | 1 year
  The modified Duke Anticoagulation Satisfaction Scale is a 14 item scale addressing the negative and positive impacts of anticoagulation with participants rating items as "strongly agree", "agree", "neither agree nor disagree", "disagree", or "strongly disagree"
Bruising using a Likert scale | 1 year
  A one item survey with the question "Over the past 3 months, have you noticed any abnormal bruising?" with response ranging from 0 (no bruising) to 10 (lots of bruising).

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Center, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Study data will be disclosed after successful conclusion of the definitive phase 3 study

REFERENCES:
- [Derived] Abdulrehman J, Forte S, Tomlinson G, Solh Z, Bolster L, Sun HL, Kuo KHM. Challenges in Trials in Sickle Cell Disease: Thromboprophylaxis in Sickle Cell Disease With Central Venous Catheters (THIS) Pilot Study. J Clin Apher. 2025 Dec;40(6):e70072. doi: 10.1002/jca.70072. PMID 41249873
- [Derived] Abdulrehman J, Forte S, Tomlinson G, Solh Z, Bolster L, Sun HL, Bartolucci P, Kuo KHM. THromboprophylaxis In Sickle Cell Disease with central venous catheters (THIS): an internal pilot randomised controlled trial protocol. BMJ Open. 2024 Jan 3;14(1):e079363. doi: 10.1136/bmjopen-2023-079363. PMID 38171625